CLINICAL TRIAL: NCT03570528
Title: Retrospective Analysis of the Differences in the Anatomy of the Nasotracheal Intubation Pathway With Computerized Tomography of Patients With Indication of Maxillary Advancement
Brief Title: CT Analysis of the Anatomy of the Nasotracheal Intubation Pathway of Patients With Indication of Maxillary Advancement
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Instructor, Ankara University
Other Study IDs: 08/03
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Maxillary Hypoplasia; Retrognathia; Intubation; Tomography
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maxillary Retrusion: CT
- Healthy Patients

SUMMARY:
Differences in nasotracheal intubation pathway anatomy will be observed between healthy patients and patients with maxillary retrusion.

The results will clarify the nasotracheal intubation tube preference for these patients.

DETAILED DESCRIPTION:
A combination of many factors affecting growth and development creates dento-facial deformities. One of these deformities may be defined as maxillary retrusion defined as inadequate maxillary development . The maxilla's sagittal skeletal deficiencies cause functional problems such as respiratory and nutritional difficulties in addition to aesthetic problems and often require surgical treatment.

These surgeries are done under general anesthesia. Nasotracheal intubation is used during these surgeries to provide general anesthesia. During nasotracheal intubation, there are two different pathways (upper and lower) in which the tracheal tube can advance through the nostrils.

The lower tract extends along the nasal floor and lies beneath the lower concha. Concha nasalis inferior is a thin and independent viscerocranium bone and articulates with the face of the maxillary and palatine bone facing the nasal cavity of the vertical lamina. The free lower edge of the concha nasalis inferior is oriented downwards towards the nasal cavity, restricting the meatus inferior. The inferior of the meatus is the largest and extends along the length of the outer wall of the nasal cavity. The area where the part between the first ⅓ and the middle ⅓ meets is the widest area of meatus nasi medius and there is the openness of the nasolacrimal channel. In the lower opening of the nasolacrimal duct, there may be an indeterminate mucosa layer formed by the mucous membrane of the nasal cavity, which is called Hasner cap.

The upper pathway is located just below the middle concha over the lower concha. Concha nasal is medius is a segment extending medially from the ethmoid bone and may sometimes contain one or more of the ethmoid air cells. Concha nasalis medius extends to the posterior and articulates with a vertical laminate of palatine bone. Below Concha nasalis medius is called meatus nasi medius and narrows from front to back. The widest area of the beginning of meatus nasi medius, just above the vestibulum, is called the atrium meatus medii. There are many paranasal sinuses in Meatus nasi medius; frontal sinus, anterior and middle group ethmoid sinuses and maxillary sinus opens here. At the extreme end of the Meatus nasi medius, there are foramen sphenopalatinum, which vessels and nerves related to the nasal cavity enter this gap.

The lower pathway is referred to as a safer road than the upper pathway, since it is located remote from the middle concha and from the cribriform layer. The trauma to the middle concha may cause avulsions and large bleedings. Trauma to the cribriform plate may also cause cerebrospinal fluid rhinoresin or olfactory nerve damage. These conditions will be especially important in anatomic variations, such as in middle concha hypertrophy and concha bullosa.

The fact that the anesthetist has knowledge of the regional anatomy and the ability to choose the appropriate size of the intubation canal is important for preventing these complications. The purpose of the current study is to study complete head tomography images for patients with maxillary retrusions and evaluate bone and soft tissue anatomy and reveal the differences which can be found in airway size and to use intubation tubes accordingly to these data.

Eight different parameters, including diameter measurements for two different intubation routes,in right / left separation, male / female separation and patient / control group separation will be evaluated.

In the study, effect size (f) = 0.275, α = 0.05, β = 0.80 and 1-and 80% at 95% confidence theoretical power for each group in this study 100 d enek is calculated. Investigators aimed to study the patient capacity of the department with a minimum of 51 patients in each group.

The data for the study will be evaluated by the licensed SPSS 21.0 package program. Student's t test and / or Mann-Whitney U test in two-group comparisons and Anova and / or Kruskall-Wallis H test in three or more group comparisons as a result of normality tests of the data. Correlation analysis or chi-square dependence tests will be used to relate variables according to the level of measurement of the data. For the intra-observer reliability, the Kap p a compliance test will be used. It should be stated that there is no significant difference when p> 0,05 and when p <0,05 meaningful difference will be indicated.

ELIGIBILITY:
Inclusion Criteria:

CT data of patients with indications for maxillary advancement surgery will be included in the study.

Exclusion Criteria:

CT images without nasal cavities will not be included in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who underwent surgery with indication of maxillary advancement.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Tube Size | 2 months
  Minimum nasotracheal tube sizes will be calculated (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)